CLINICAL TRIAL: NCT05593055
Title: Mineralocorticoid Receptor, Coronary Microvascular Function, and Cardiac Efficiency in Hypertension
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gail Kurr Adler, Chief, Cardiovascular Endocrinology Section, Principal Investigator, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2022P002126
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Left Ventricular Hypertrophy
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular | interventions — Eplerenone; Chlorthalidone; Potassium

STUDY DESIGN:
Intervention Model Description: Participants are randomized to chlorthalidone or eplerenone.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eplerenone (Active Comparator): Participants be placed on enalapril 10 mg and weaned off their other anti-hypertensives prior to the Pre-Treatment Assessment. Amlodipine (5 to 10 mg) will be added if needed to control blood pressure. After the Pre-Treatment Assessment, participants randomized to this arm will receive 50 mg eplerenone . At 2 weeks, eplerenone will be increased to 100 mg. Amlodipine (5 to 10 mg) will be added at 6 weeks or later if needed to achieve the BP target of <135/85 mmHg.
  Interventions: Drug: Eplerenone
- Chlorthalidone + potassium (Active Comparator): Participants be placed on enalapril 10 mg and weaned off their other anti-hypertensives prior to the Pre-Treatment Assessment. Amlodipine (5 to 10 mg) will be added if needed to control blood pressure. After the Pre-Treatment Assessment, participants randomized to this arm will receive 12.5 mg chlorthalidone + 10 mEq potassium. At 2 weeks, chlorthalidone will be increased to 25 mg + 20 mEq potassium. Amlodipine (5 to 10 mg) will be added at 6 weeks or later if needed to achieve the BP target of <135/85 mmHg.
  Interventions: Drug: Chlorthalidone; Drug: Potassium

INTERVENTIONS:
Drug: Eplerenone — After the Pre-Treatment Assessment, participants in the eplerenone arm will be given 50 mg eplerenone. At 2 weeks, eplerenone will be increased to 100 mg.
  Arms: Eplerenone
Drug: Chlorthalidone — After the Pre-Treatment Assessment, participants in the chlorthalidone arm will be given 12.5 mg chlorthalidone + 10 mEq potassium. At 2 weeks, chlorthalidone will be increased to 25 mg + 20 mEq potassium.
  Arms: Chlorthalidone + potassium
Drug: Potassium — After the Pre-Treatment Assessment, participants in the chlorthalidone arm will be given 12.5 mg chlorthalidone + 10 mEq potassium. At 2 weeks, chlorthalidone will be increased to 25 mg + 20 mEq potassium.
  Arms: Chlorthalidone + potassium

SUMMARY:
The investigators' goal is to show that in hypertensive men and women with left ventricular hypertrophy (LVH) treatment with a mineralocorticoid receptor (MR) antagonist, versus a thiazide-like diuretic, will improve coronary microvascular function and cardiac efficiency, which will associate with improvements in LV structure and function. The investigators will achieve this through a randomized, controlled, basic experimental study involving humans (BESH).

DETAILED DESCRIPTION:
The investigators are recruiting individuals with hypertension and LVH, as defined by echocardiography, who are on chronic angiotensin converting enzyme inhibitor (ACEi) or angiotensin receptor blockade (ARB). Participants will be transitioned to enalapril, ACEi, with washout of all other anti-hypertensives and then randomized to add-on treatment for 9 months with eplerenone (MR antagonist) or chlorthalidone (thiazide-like diuretic) + potassium. The investigators will use cardiac PET to quantify changes in coronary microvascular function and cardiac efficiency; echocardiography to assess changes in cardiac function and structure. The investigators will define the impact of eplerenone as compared with chlorthalidone on coronary microvascular function (Aim 1) and cardiac efficiency (Aim 2) and determine the relationship between coronary microvascular function and cardiac efficiency. Additionally, the investigators will determine whether improvements in coronary microvascular function and/or cardiac efficiency correlate with improvements in myocardial structure and function (chamber dimensions, diastolic function, and global longitudinal strain) in individuals with hypertension and LVH.

Participants be placed on enalapril 10 mg and weaned off their other anti-hypertensives prior to the Pre-Treatment Assessment. After the Pre-Treatment Assessment, participants will be randomized to the following daily medications: 50 mg eplerenone or 12.5 mg chlorthalidone + 10 mEq potassium. At 2 weeks, eplerenone will be increased to 100 mg and chlorthalidone to 25 mg + 20 mEq potassium. Amlodipine (5 to 10 mg) will be added at 6 weeks or later if needed to achieve the BP target of <135/85 mmHg. Study outcomes will be assessed at baseline and 9 months after randomization. The primary outcome measures will be: 1) myocardial flow reserve (MFR, ratio of stress over rest myocardial blood flow); and 2) myocardial external efficiency (MEE, ratio of myocardial work over myocardial oxygen consumption and LV mass). The investigators will also measure: 1) myocardial oxygen consumption (MVO2); 2) myocardial function (peak global longitudinal strain, tissue Doppler mitral annular early diastolic relaxation velocity [e'], and the ratio of mitral E velocity to e' [E/e']) as measured by 2D echocardiography; 3) markers of cardiovascular injury and remodeling, including high sensitivity troponin and procollagen III amino terminal propeptide (PIIINP); and 4) measures of renin-angiotensin-aldosterone system under resting conditions, with upright posture, and with angiotensin-II stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. History of hypertension

   1. Seated systolic BP < 180 mmHg and diastolic < 110 mmHg if on antihypertensives
   2. Seated systolic BP 141-200 mmHg and/or diastolic BP 90-114 mmHg if not on antihypertensives
2. LVH by echocardiogram

   1. For men: interventricular septum thickness ≥ 12mm
   2. For women: interventricular septum thickness ≥ 11mm
3. We will also allow inclusion of people with treated hypothyroidism, pre-diabetes and diabetes controlled by diet, exercise, and/or metformin.

Exclusion Criteria:

* Use of MR antagonist (eplerenone, spironolactone, or finerenone) or amiloride (amiloride inhibits ENaC, which is a key mediator of MR's actions) within the past year
* Orthostatic hypotension
* Major medical illness, including uncontrolled diabetes mellitus (Hemoglobin A1c >7.5)
* LV ejection fraction < 40%
* New York Heart Association class III to IV congestive heart failure or unstable angina
* A history in the prior 6 months of Q-wave myocardial infarction, stroke, transient ischemic attack, percutaneous transluminal coronary angioplasty, or coronary artery bypass graft
* History of secondary hypertension
* Known genetic cardiomyopathy
* Renal disease (seum creatinine >1.5 mg/dL for men and >1.3 mg/dL for women)
* Hepatic disease
* Bronchospastic lung disease
* Alcohol or substance abuse
* Hormone replacement therapy
* Abnormal values for electrolytes, liver enzymes or TSH
* Pregnancy or lactation
* All individuals <18 and >75 years will be excluded due to safety concerns of administering an angiotensin-II infusion in these patient groups.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in myocardial flow reserve | 9 months
  Change in myocardial flow reserve (ratio of hyperemic stress myocardial blood flow to rest myocardial blood flow)

SECONDARY OUTCOMES:
Change in myocardial external efficiency | 9 months
  Change in myocardial external efficiency (ratio of myocardial work to oxygen consumption)

CONTACTS AND LOCATIONS:
Overall Officials: Gail K Adler, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Johnson K, Oparil S, Davis BR, Tereshchenko LG. Prevention of Heart Failure in Hypertension-Disentangling the Role of Evolving Left Ventricular Hypertrophy and Blood Pressure Lowering: The ALLHAT Study. J Am Heart Assoc. 2019 Apr 16;8(8):e011961. doi: 10.1161/JAHA.119.011961. PMID 30943832
- [Background] Jaffe IZ, Mendelsohn ME. Angiotensin II and aldosterone regulate gene transcription via functional mineralocortocoid receptors in human coronary artery smooth muscle cells. Circ Res. 2005 Apr 1;96(6):643-50. doi: 10.1161/01.RES.0000159937.05502.d1. Epub 2005 Feb 17. PMID 15718497
- [Background] Luther JM, Luo P, Wang Z, Cohen SE, Kim HS, Fogo AB, Brown NJ. Aldosterone deficiency and mineralocorticoid receptor antagonism prevent angiotensin II-induced cardiac, renal, and vascular injury. Kidney Int. 2012 Sep;82(6):643-51. doi: 10.1038/ki.2012.170. Epub 2012 May 23. PMID 22622494
- [Background] DeMarco VG, Habibi J, Jia G, Aroor AR, Ramirez-Perez FI, Martinez-Lemus LA, Bender SB, Garro M, Hayden MR, Sun Z, Meininger GA, Manrique C, Whaley-Connell A, Sowers JR. Low-Dose Mineralocorticoid Receptor Blockade Prevents Western Diet-Induced Arterial Stiffening in Female Mice. Hypertension. 2015 Jul;66(1):99-107. doi: 10.1161/HYPERTENSIONAHA.115.05674. Epub 2015 May 26. PMID 26015449
- [Background] Galmiche G, Pizard A, Gueret A, El Moghrabi S, Ouvrard-Pascaud A, Berger S, Challande P, Jaffe IZ, Labat C, Lacolley P, Jaisser F. Smooth muscle cell mineralocorticoid receptors are mandatory for aldosterone-salt to induce vascular stiffness. Hypertension. 2014 Mar;63(3):520-526. doi: 10.1161/HYPERTENSIONAHA.113.01967. Epub 2013 Dec 2. PMID 24296280
- [Background] Schiffrin EL. Effects of aldosterone on the vasculature. Hypertension. 2006 Mar;47(3):312-8. doi: 10.1161/01.HYP.0000201443.63240.a7. Epub 2006 Jan 23. No abstract available. PMID 16432039
- [Background] Maron BA, Leopold JA. Mineralocorticoid receptor antagonists and endothelial function. Curr Opin Investig Drugs. 2008 Sep;9(9):963-9. PMID 18729003
- [Background] Lieb W, Larson MG, Benjamin EJ, Yin X, Tofler GH, Selhub J, Jacques PF, Wang TJ, Vita JA, Levy D, Vasan RS, Mitchell GF. Multimarker approach to evaluate correlates of vascular stiffness: the Framingham Heart Study. Circulation. 2009 Jan 6;119(1):37-43. doi: 10.1161/CIRCULATIONAHA.108.816108. Epub 2008 Dec 22. PMID 19103986
- [Background] Connell JM, MacKenzie SM, Freel EM, Fraser R, Davies E. A lifetime of aldosterone excess: long-term consequences of altered regulation of aldosterone production for cardiovascular function. Endocr Rev. 2008 Apr;29(2):133-54. doi: 10.1210/er.2007-0030. Epub 2008 Feb 21. PMID 18292466
- [Background] Pitt B, Reichek N, Willenbrock R, Zannad F, Phillips RA, Roniker B, Kleiman J, Krause S, Burns D, Williams GH. Effects of eplerenone, enalapril, and eplerenone/enalapril in patients with essential hypertension and left ventricular hypertrophy: the 4E-left ventricular hypertrophy study. Circulation. 2003 Oct 14;108(15):1831-8. doi: 10.1161/01.CIR.0000091405.00772.6E. Epub 2003 Sep 29. PMID 14517164
- [Background] Pitt B, Zannad F, Remme WJ, Cody R, Castaigne A, Perez A, Palensky J, Wittes J. The effect of spironolactone on morbidity and mortality in patients with severe heart failure. Randomized Aldactone Evaluation Study Investigators. N Engl J Med. 1999 Sep 2;341(10):709-17. doi: 10.1056/NEJM199909023411001. PMID 10471456
- [Background] Pitt B, Remme W, Zannad F, Neaton J, Martinez F, Roniker B, Bittman R, Hurley S, Kleiman J, Gatlin M; Eplerenone Post-Acute Myocardial Infarction Heart Failure Efficacy and Survival Study Investigators. Eplerenone, a selective aldosterone blocker, in patients with left ventricular dysfunction after myocardial infarction. N Engl J Med. 2003 Apr 3;348(14):1309-21. doi: 10.1056/NEJMoa030207. Epub 2003 Mar 31. PMID 12668699
- [Background] Zannad F, McMurray JJ, Krum H, van Veldhuisen DJ, Swedberg K, Shi H, Vincent J, Pocock SJ, Pitt B; EMPHASIS-HF Study Group. Eplerenone in patients with systolic heart failure and mild symptoms. N Engl J Med. 2011 Jan 6;364(1):11-21. doi: 10.1056/NEJMoa1009492. Epub 2010 Nov 14. PMID 21073363
- [Background] Bakris GL, Agarwal R, Anker SD, Pitt B, Ruilope LM, Rossing P, Kolkhof P, Nowack C, Schloemer P, Joseph A, Filippatos G; FIDELIO-DKD Investigators. Effect of Finerenone on Chronic Kidney Disease Outcomes in Type 2 Diabetes. N Engl J Med. 2020 Dec 3;383(23):2219-2229. doi: 10.1056/NEJMoa2025845. Epub 2020 Oct 23. PMID 33264825
- [Background] Filippatos G, Anker SD, Agarwal R, Pitt B, Ruilope LM, Rossing P, Kolkhof P, Schloemer P, Tornus I, Joseph A, Bakris GL; FIDELIO-DKD Investigators. Finerenone and Cardiovascular Outcomes in Patients With Chronic Kidney Disease and Type 2 Diabetes. Circulation. 2021 Feb 9;143(6):540-552. doi: 10.1161/CIRCULATIONAHA.120.051898. Epub 2020 Nov 16. PMID 33198491
- [Background] Zhou W, Brown JM, Bajaj NS, Chandra A, Divakaran S, Weber B, Bibbo CF, Hainer J, Taqueti VR, Dorbala S, Blankstein R, Adler D, O'Gara P, Di Carli MF. Hypertensive coronary microvascular dysfunction: a subclinical marker of end organ damage and heart failure. Eur Heart J. 2020 Jul 1;41(25):2366-2375. doi: 10.1093/eurheartj/ehaa191. PMID 32221588
- [Background] Bajaj NS, Singh A, Zhou W, Gupta A, Fujikura K, Byrne C, Harms HJ, Osborne MT, Bravo P, Andrikopolou E, Divakaran S, Bibbo CF, Hainer J, Skali H, Taqueti V, Steigner M, Dorbala S, Charytan DM, Prabhu SD, Blankstein R, Deo RC, Solomon SD, Di Carli MF. Coronary Microvascular Dysfunction, Left Ventricular Remodeling, and Clinical Outcomes in Patients With Chronic Kidney Impairment. Circulation. 2020 Jan 7;141(1):21-33. doi: 10.1161/CIRCULATIONAHA.119.043916. Epub 2019 Nov 29. PMID 31779467
- [Background] Taqueti VR, Solomon SD, Shah AM, Desai AS, Groarke JD, Osborne MT, Hainer J, Bibbo CF, Dorbala S, Blankstein R, Di Carli MF. Coronary microvascular dysfunction and future risk of heart failure with preserved ejection fraction. Eur Heart J. 2018 Mar 7;39(10):840-849. doi: 10.1093/eurheartj/ehx721. PMID 29293969
- [Background] Camici PG, Crea F. Coronary microvascular dysfunction. N Engl J Med. 2007 Feb 22;356(8):830-40. doi: 10.1056/NEJMra061889. No abstract available. PMID 17314342
- [Background] Prior JO, Quinones MJ, Hernandez-Pampaloni M, Facta AD, Schindler TH, Sayre JW, Hsueh WA, Schelbert HR. Coronary circulatory dysfunction in insulin resistance, impaired glucose tolerance, and type 2 diabetes mellitus. Circulation. 2005 May 10;111(18):2291-8. doi: 10.1161/01.CIR.0000164232.62768.51. Epub 2005 Apr 25. PMID 15851590
- [Background] Brush JE Jr, Cannon RO 3rd, Schenke WH, Bonow RO, Leon MB, Maron BJ, Epstein SE. Angina due to coronary microvascular disease in hypertensive patients without left ventricular hypertrophy. N Engl J Med. 1988 Nov 17;319(20):1302-7. doi: 10.1056/NEJM198811173192002. PMID 3185633
- [Background] Opherk D, Mall G, Zebe H, Schwarz F, Weihe E, Manthey J, Kubler W. Reduction of coronary reserve: a mechanism for angina pectoris in patients with arterial hypertension and normal coronary arteries. Circulation. 1984 Jan;69(1):1-7. doi: 10.1161/01.cir.69.1.1. PMID 6689632
- [Background] Hamasaki S, Al Suwaidi J, Higano ST, Miyauchi K, Holmes DR Jr, Lerman A. Attenuated coronary flow reserve and vascular remodeling in patients with hypertension and left ventricular hypertrophy. J Am Coll Cardiol. 2000 May;35(6):1654-60. doi: 10.1016/s0735-1097(00)00594-5. PMID 10807473
- [Background] Garg R, Rao AD, Baimas-George M, Hurwitz S, Foster C, Shah RV, Jerosch-Herold M, Kwong RY, Di Carli MF, Adler GK. Mineralocorticoid receptor blockade improves coronary microvascular function in individuals with type 2 diabetes. Diabetes. 2015 Jan;64(1):236-42. doi: 10.2337/db14-0670. Epub 2014 Aug 14. PMID 25125488
- [Background] Kim SK, Biwer LA, Moss ME, Man JJ, Aronovitz MJ, Martin GL, Carrillo-Salinas FJ, Salvador AM, Alcaide P, Jaffe IZ. Mineralocorticoid Receptor in Smooth Muscle Contributes to Pressure Overload-Induced Heart Failure. Circ Heart Fail. 2021 Feb;14(2):e007279. doi: 10.1161/CIRCHEARTFAILURE.120.007279. Epub 2021 Feb 1. PMID 33517669
- [Background] Rocha R, Stier CT Jr, Kifor I, Ochoa-Maya MR, Rennke HG, Williams GH, Adler GK. Aldosterone: a mediator of myocardial necrosis and renal arteriopathy. Endocrinology. 2000 Oct;141(10):3871-8. doi: 10.1210/endo.141.10.7711. PMID 11014244
- [Background] Oestreicher EM, Martinez-Vasquez D, Stone JR, Jonasson L, Roubsanthisuk W, Mukasa K, Adler GK. Aldosterone and not plasminogen activator inhibitor-1 is a critical mediator of early angiotensin II/NG-nitro-L-arginine methyl ester-induced myocardial injury. Circulation. 2003 Nov 18;108(20):2517-23. doi: 10.1161/01.CIR.0000097000.51723.6F. Epub 2003 Oct 27. PMID 14581407
- [Background] Bender SB, DeMarco VG, Padilla J, Jenkins NT, Habibi J, Garro M, Pulakat L, Aroor AR, Jaffe IZ, Sowers JR. Mineralocorticoid receptor antagonism treats obesity-associated cardiac diastolic dysfunction. Hypertension. 2015 May;65(5):1082-8. doi: 10.1161/HYPERTENSIONAHA.114.04912. Epub 2015 Feb 23. PMID 25712719
- [Background] Mueller KB, Bender SB, Hong K, Yang Y, Aronovitz M, Jaisser F, Hill MA, Jaffe IZ. Endothelial Mineralocorticoid Receptors Differentially Contribute to Coronary and Mesenteric Vascular Function Without Modulating Blood Pressure. Hypertension. 2015 Nov;66(5):988-97. doi: 10.1161/HYPERTENSIONAHA.115.06172. Epub 2015 Sep 8. PMID 26351033
- [Background] Sorensen J, Harms HJ, Aalen JM, Baron T, Smiseth OA, Flachskampf FA. Myocardial Efficiency: A Fundamental Physiological Concept on the Verge of Clinical Impact. JACC Cardiovasc Imaging. 2020 Jul;13(7):1564-1576. doi: 10.1016/j.jcmg.2019.08.030. Epub 2019 Dec 18. PMID 31864979
- [Background] Brown DA, Perry JB, Allen ME, Sabbah HN, Stauffer BL, Shaikh SR, Cleland JG, Colucci WS, Butler J, Voors AA, Anker SD, Pitt B, Pieske B, Filippatos G, Greene SJ, Gheorghiade M. Expert consensus document: Mitochondrial function as a therapeutic target in heart failure. Nat Rev Cardiol. 2017 Apr;14(4):238-250. doi: 10.1038/nrcardio.2016.203. Epub 2016 Dec 22. PMID 28004807
- [Background] Zhou B, Tian R. Mitochondrial dysfunction in pathophysiology of heart failure. J Clin Invest. 2018 Aug 31;128(9):3716-3726. doi: 10.1172/JCI120849. Epub 2018 Aug 20. PMID 30124471
- [Background] Hafstad AD, Nabeebaccus AA, Shah AM. Novel aspects of ROS signalling in heart failure. Basic Res Cardiol. 2013 Jul;108(4):359. doi: 10.1007/s00395-013-0359-8. Epub 2013 Jun 6. PMID 23740217
- [Background] Peterson LR, Herrero P, Schechtman KB, Racette SB, Waggoner AD, Kisrieva-Ware Z, Dence C, Klein S, Marsala J, Meyer T, Gropler RJ. Effect of obesity and insulin resistance on myocardial substrate metabolism and efficiency in young women. Circulation. 2004 May 11;109(18):2191-6. doi: 10.1161/01.CIR.0000127959.28627.F8. Epub 2004 May 3. PMID 15123530
- [Background] Mazumder PK, O'Neill BT, Roberts MW, Buchanan J, Yun UJ, Cooksey RC, Boudina S, Abel ED. Impaired cardiac efficiency and increased fatty acid oxidation in insulin-resistant ob/ob mouse hearts. Diabetes. 2004 Sep;53(9):2366-74. doi: 10.2337/diabetes.53.9.2366. PMID 15331547
- [Background] Boudina S, Sena S, O'Neill BT, Tathireddy P, Young ME, Abel ED. Reduced mitochondrial oxidative capacity and increased mitochondrial uncoupling impair myocardial energetics in obesity. Circulation. 2005 Oct 25;112(17):2686-95. doi: 10.1161/CIRCULATIONAHA.105.554360. PMID 16246967
- [Background] How OJ, Aasum E, Severson DL, Chan WY, Essop MF, Larsen TS. Increased myocardial oxygen consumption reduces cardiac efficiency in diabetic mice. Diabetes. 2006 Feb;55(2):466-73. doi: 10.2337/diabetes.55.02.06.db05-1164. PMID 16443782
- [Background] Buchanan J, Mazumder PK, Hu P, Chakrabarti G, Roberts MW, Yun UJ, Cooksey RC, Litwin SE, Abel ED. Reduced cardiac efficiency and altered substrate metabolism precedes the onset of hyperglycemia and contractile dysfunction in two mouse models of insulin resistance and obesity. Endocrinology. 2005 Dec;146(12):5341-9. doi: 10.1210/en.2005-0938. Epub 2005 Sep 1. PMID 16141388
- [Background] Laine H, Katoh C, Luotolahti M, Yki-Jarvinen H, Kantola I, Jula A, Takala TO, Ruotsalainen U, Iida H, Haaparanta M, Nuutila P, Knuuti J. Myocardial oxygen consumption is unchanged but efficiency is reduced in patients with essential hypertension and left ventricular hypertrophy. Circulation. 1999 Dec 14;100(24):2425-30. doi: 10.1161/01.cir.100.24.2425. PMID 10595955
- [Background] Kim IS, Izawa H, Sobue T, Ishihara H, Somura F, Nishizawa T, Nagata K, Iwase M, Yokota M. Prognostic value of mechanical efficiency in ambulatory patients with idiopathic dilated cardiomyopathy in sinus rhythm. J Am Coll Cardiol. 2002 Apr 17;39(8):1264-8. doi: 10.1016/s0735-1097(02)01775-8. PMID 11955842
- [Background] Beanlands RS, Nahmias C, Gordon E, Coates G, deKemp R, Firnau G, Fallen E. The effects of beta(1)-blockade on oxidative metabolism and the metabolic cost of ventricular work in patients with left ventricular dysfunction: A double-blind, placebo-controlled, positron-emission tomography study. Circulation. 2000 Oct 24;102(17):2070-5. doi: 10.1161/01.cir.102.17.2070. PMID 11044422
- [Background] Hung CS (啟盛) 628401, Chang YY, Tsai CH, Liao CW, Peng SY, Lee BC, Pan CT, Wu XM, Chen ZW, Wu VC, Wan CH, Young MJ, Chou CH, Lin YH; TAIPAI Study Group. Aldosterone suppresses cardiac mitochondria. Transl Res. 2022 Jan;239:58-70. doi: 10.1016/j.trsl.2021.08.003. Epub 2021 Aug 16. PMID 34411778
- [Background] Tsai CH, Pan CT, Chang YY, Peng SY, Lee PC, Liao CW, Shun CT, Li PT, Wu VC, Chou CH, Tsai IJ, Hung CS, Lin YH. Aldosterone Excess Induced Mitochondria Decrease and Dysfunction via Mineralocorticoid Receptor and Oxidative Stress In Vitro and In Vivo. Biomedicines. 2021 Aug 2;9(8):946. doi: 10.3390/biomedicines9080946. PMID 34440149
- [Background] Ibarrola J, Sadaba R, Martinez-Martinez E, Garcia-Pena A, Arrieta V, Alvarez V, Fernandez-Celis A, Gainza A, Cachofeiro V, Santamaria E, Fernandez-Irigoyen J, Jaisser F, Lopez-Andres N. Aldosterone Impairs Mitochondrial Function in Human Cardiac Fibroblasts via A-Kinase Anchor Protein 12. Sci Rep. 2018 May 1;8(1):6801. doi: 10.1038/s41598-018-25068-6. PMID 29717226
- [Background] Bell SP, Adkisson DW, Lawson MA, Wang L, Ooi H, Sawyer DB, Kronenberg MW. Antifailure therapy including spironolactone improves left ventricular energy supply-demand relations in nonischemic dilated cardiomyopathy. J Am Heart Assoc. 2014 Aug 27;3(4):e000883. doi: 10.1161/JAHA.114.000883. PMID 25164945
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2018 May 15;71(19):e127-e248. doi: 10.1016/j.jacc.2017.11.006. Epub 2017 Nov 13. No abstract available. PMID 29146535
- [Background] Epstein M, Williams GH, Weinberger M, Lewin A, Krause S, Mukherjee R, Patni R, Beckerman B. Selective aldosterone blockade with eplerenone reduces albuminuria in patients with type 2 diabetes. Clin J Am Soc Nephrol. 2006 Sep;1(5):940-51. doi: 10.2215/CJN.00240106. Epub 2006 Jul 19. PMID 17699311
- [Background] Cushman WC, Ford CE, Cutler JA, Margolis KL, Davis BR, Grimm RH, Black HR, Hamilton BP, Holland J, Nwachuku C, Papademetriou V, Probstfield J, Wright JT Jr, Alderman MH, Weiss RJ, Piller L, Bettencourt J, Walsh SM; ALLHAT Collaborative Research Group. Success and predictors of blood pressure control in diverse North American settings: the antihypertensive and lipid-lowering treatment to prevent heart attack trial (ALLHAT). J Clin Hypertens (Greenwich). 2002 Nov-Dec;4(6):393-404. doi: 10.1111/j.1524-6175.2002.02045.x. PMID 12461301
- [Background] Olde Engberink RH, Frenkel WJ, van den Bogaard B, Brewster LM, Vogt L, van den Born BJ. Effects of thiazide-type and thiazide-like diuretics on cardiovascular events and mortality: systematic review and meta-analysis. Hypertension. 2015 May;65(5):1033-40. doi: 10.1161/HYPERTENSIONAHA.114.05122. Epub 2015 Mar 2. PMID 25733241
- [Background] Stone IB, Green JAEM, Koefoed AW, Hornik ES, Williams JS, Adler GK, Williams GH. Striatin genotype-based, mineralocorticoid receptor antagonist-driven clinical trial: study rationale and design. Pharmacogenet Genomics. 2021 Jun 1;31(4):83-88. doi: 10.1097/FPC.0000000000000425. PMID 33904521
- [Background] Raji A, Williams GH, Jeunemaitre X, Hopkins PN, Hunt SC, Hollenberg NK, Seely EW. Insulin resistance in hypertensives: effect of salt sensitivity, renin status and sodium intake. J Hypertens. 2001 Jan;19(1):99-105. doi: 10.1097/00004872-200101000-00013. PMID 11204310
- [Background] Chamarthi B, Williams JS, Williams GH. A mechanism for salt-sensitive hypertension: abnormal dietary sodium-mediated vascular response to angiotensin-II. J Hypertens. 2010 May;28(5):1020-6. doi: 10.1097/HJH.0b013e3283375974. PMID 20216091
- [Background] Pojoga L, Kolatkar NS, Williams JS, Perlstein TS, Jeunemaitre X, Brown NJ, Hopkins PN, Raby BA, Williams GH. Beta-2 adrenergic receptor diplotype defines a subset of salt-sensitive hypertension. Hypertension. 2006 Nov;48(5):892-900. doi: 10.1161/01.HYP.0000244688.45472.95. Epub 2006 Oct 2. PMID 17015767
- [Background] Underwood PC, Sun B, Williams JS, Pojoga LH, Chamarthi B, Lasky-Su J, Raby BA, Hopkins PN, Jeunemaitre X, Brown NJ, Adler GK, Williams GH. The relationship between peroxisome proliferator-activated receptor-gamma and renin: a human genetics study. J Clin Endocrinol Metab. 2010 Sep;95(9):E75-9. doi: 10.1210/jc.2010-0270. Epub 2010 Jul 14. PMID 20631015
- [Background] Bentley-Lewis R, Adler GK, Perlstein T, Seely EW, Hopkins PN, Williams GH, Garg R. Body mass index predicts aldosterone production in normotensive adults on a high-salt diet. J Clin Endocrinol Metab. 2007 Nov;92(11):4472-5. doi: 10.1210/jc.2007-1088. Epub 2007 Aug 28. PMID 17726083
- [Background] Baudrand R, Pojoga LH, Vaidya A, Garza AE, Vohringer PA, Jeunemaitre X, Hopkins PN, Yao TM, Williams J, Adler GK, Williams GH. Statin Use and Adrenal Aldosterone Production in Hypertensive and Diabetic Subjects. Circulation. 2015 Nov 10;132(19):1825-33. doi: 10.1161/CIRCULATIONAHA.115.016759. Epub 2015 Oct 2. PMID 26432671
- [Background] Haas AV, Baudrand R, Easly RM, Murray GR, Touyz RM, Pojoga LH, Jeunemaitre X, Hopkins PN, Rosner B, Williams JS, Williams GH, Adler GK. Interplay Between Statins, Cav1 (Caveolin-1), and Aldosterone. Hypertension. 2020 Sep;76(3):962-967. doi: 10.1161/HYPERTENSIONAHA.120.14777. Epub 2020 Aug 3. PMID 32755411
- [Background] Hollenberg NK, Chenitz WR, Adams DF, Williams GH. Reciprocal influence of salt intake on adrenal glomerulosa and renal vascular responses to angiotensin II in normal man. J Clin Invest. 1974 Jul;54(1):34-42. doi: 10.1172/JCI107748. PMID 4365595
- [Background] Harnack LJ, Cogswell ME, Shikany JM, Gardner CD, Gillespie C, Loria CM, Zhou X, Yuan K, Steffen LM. Sources of Sodium in US Adults From 3 Geographic Regions. Circulation. 2017 May 9;135(19):1775-1783. doi: 10.1161/CIRCULATIONAHA.116.024446. PMID 28483828